CLINICAL TRIAL: NCT04732468
Title: Phase 1b Open-Label Study of the Safety, Reactogenicity, and Immunogenicity of Subcutaneously and Orally Administered Prophylactic Vaccination With 2nd Generation (E1/E2B/E3-Deleted) Adenoviral COVID-19 in Normal Healthy Volunteers
Brief Title: COVID-19 Oral and Subcutaneous Vaccination Using a 2nd Generation (E1/E2B/E3-Deleted) Adenovirus Platform in Healthy Volunteers in USA
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: The study was terminated early due to low enrollment.
Sponsor: ImmunityBio, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: COVID-4.005
Record Dates: First submitted 2021-01-27; First posted 2021-02-01 (Actual); Results first posted 2024-10-15 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-09

CONDITIONS: Covid19
MeSH Terms: conditions — COVID-19 | interventions — Suspensions; Injections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Cohort 1- hAd5-S-Fusion+N-ETSD (Suspension for injection) and hAd5-SFusion+ N-ETSD (Oral capsule) (Experimental): For subjects in cohort 1, hAd5-S-Fusion+N-ETSD (Suspension for injection) and hAd5-SFusion+N-ETSD (Oral capsule) were administered on day 1 (prime) and hAd5-S-Fusion+N-ETSD (Suspension for injection) again on day 22 (boost).
  Interventions: Biological: hAd5-S-Fusion+N-ETSD (Suspension for injection); Drug: hAd5-SFusion+ N-ETSD (Oral capsule)
- Cohort 2- hAd5-S-Fusion+N-ETSD (Suspension for injection) and hAd5-SFusion+ N-ETSD (Oral capsule) (Experimental): For subjects in cohort 2, hAd5-S-Fusion+N-ETSD (Suspension for injection) and hAd5-SFusion+N-ETSD (Oral capsule) were administered on day 1 (prime) and hAd5-S-Fusion+N-ETSD (Oral capsule) on day 22 (boost).
  Interventions: Biological: hAd5-S-Fusion+N-ETSD (Suspension for injection); Drug: hAd5-SFusion+ N-ETSD (Oral capsule)
- Cohort 3 - hAd5-S-Fusion+N-ETSD (Oral capsule) (Experimental): For subjects in cohort 3, hAd5-S-Fusion+N-ETSD (Oral capsule) were administered on days 1 (prime) and on day 22 (boost).
  Interventions: Drug: hAd5-SFusion+ N-ETSD (Oral capsule)
- Cohort 4 - hAd5-S-Fusion+N-ETSD (Suspension for injection) and hAd5-S-Fusion+N-ETSD (Oral capsule) (Experimental): For subjects in cohort 4, hAd5-S-Fusion+N-ETSD (Suspension for injection) and hAd5-S-Fusion+N-ETSD (Oral capsule) were administered on day 1 (prime) and hAd5-SFusion+N-ETSD (Oral capsule) will be administered on days 15 (boost) and 22 (boost).
  Interventions: Biological: hAd5-S-Fusion+N-ETSD (Suspension for injection); Drug: hAd5-SFusion+ N-ETSD (Oral capsule)

INTERVENTIONS:
Biological: hAd5-S-Fusion+N-ETSD (Suspension for injection) — The hAd5-S-Fusion+N-ETSD Vaccine is a human adenovirus serotype 5 (hAd5) vector with E1/E2b/E3 deletions expressing SARS-CoV-2 viral antigen spike fusion protein and nucleocapsid with an enhanced T-cell stimulation domain.
  Arms: Cohort 1- hAd5-S-Fusion+N-ETSD (Suspension for injection) and hAd5-SFusion+ N-ETSD (Oral capsule); Cohort 2- hAd5-S-Fusion+N-ETSD (Suspension for injection) and hAd5-SFusion+ N-ETSD (Oral capsule); Cohort 4 - hAd5-S-Fusion+N-ETSD (Suspension for injection) and hAd5-S-Fusion+N-ETSD (Oral capsule)
Drug: hAd5-SFusion+ N-ETSD (Oral capsule) — The hAd5-S-Fusion+N-ETSD Vaccine is a human adenovirus serotype 5 (hAd5) vector with E1/E2b/E3 deletions expressing SARS-CoV-2 viral antigen spike fusion protein and nucleocapsid with an enhanced T-cell stimulation domain.

SUMMARY:
This is a phase 1b, open-label study in adult healthy subjects. This clinical trial is designed to assess the safety, reactogenicity, and immunogenicity the combination of hAd5-S-Fusion+N-ETSD (Suspension for injection) and hAd5-S-Fusion+N-ETSD (Oral capsule) and to select an optimal combination dose for future studies.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy adults, age 18 - 55 years, inclusive, at time of enrollment.
2. Able to understand and provide a signed informed consent that fulfills the relevant Institutional Review Board (IRB) or Independent Ethics Committee (IEC) guidelines.
3. Agrees to the collection of biospecimens (eg, nasopharyngeal [NP] swabs) and venous blood per protocol.
4. Ability to attend required study visits and return for adequate follow-up, as required by this protocol.
5. Ability to swallow a capsule.
6. Temperature < 38°C.
7. Negative for SARS-CoV-2 (qPCR or LAMP test) and no known previous COVID-19 exposure or disease.
8. Agreement to practice effective contraception for female subjects of childbearing potential and non-sterile males. Female subjects of childbearing potential must agree to use effective contraception while on study until at least 1 month after the last dose of vaccine. Non-sterile male subjects must agree to use a condom while on study until at least 1 month after the last dose of vaccine. Effective contraception includes surgical sterilization (eg, vasectomy, tubal ligation), two forms of barrier methods (eg, condom, diaphragm) used with spermicide, intrauterine devices (IUDs), oral contraceptives, and abstinence.

Exclusion Criteria:

1. Allergy to any component of the investigational vaccine, or a more severe allergic reaction and history of allergies in the past.
2. Pregnant and nursing women. A negative serum or urine pregnancy test during screening and on the day of and prior to each dose must be documented before the vaccine is administered to a female subject of childbearing potential.
3. Live in a nursing home or long-term care facility.
4. Chronic lung disease including chronic obstructive pulmonary disease (COPD) or moderate to severe asthma.
5. Pulmonary fibrosis.
6. Current or former smoker.
7. Bone marrow or organ transplantation.
8. Obesity (defined as body mass index [BMI] of 30 kg/m2 or higher).
9. Diabetes.
10. Chronic kidney disease.
11. Liver disease.
12. Sickle cell disease.
13. Thalassemia.
14. Doctors, nurses, first responders, and other healthcare workers working in direct contact with COVID-19 patients.
15. Any disease associated with acute fever, or any infection.
16. Self-reported history of severe acute respiratory syndrome (SARS).
17. History of hepatitis B or hepatitis C.
18. HIV or other acquired or hereditary immunodeficiency.
19. Serious cardiovascular diseases, such as heart failure, coronary artery disease, cardiomyopathies, arrhythmia, conduction block, myocardial infarction, pulmonary hypertension, severe hypertension without controllable drugs, etc.
20. Cerebrovascular disease.
21. Cystic fibrosis.
22. Neurologic conditions, such as dementia.
23. Hereditary or acquired angioneurotic edema.
24. Urticaria in the last 12 months.
25. No spleen or functional asplenia.
26. Platelet disorder or other bleeding disorder that may cause injection contraindication.
27. Chronic use (more than 14 continuous days) of any medications that may be associated with impaired immune responsiveness within 3 months before administration of study vaccine. (Including, but not limited to, systemic corticosteroids exceeding 10 mg/day of prednisone equivalent, allergy injections, immunoglobulin, interferon, immunomodulators. The use of low dose topical, ophthalmic, inhaled and intranasal steroid preparations will be permitted.)
28. Prior administration of blood products in last 4 months.
29. Prior administration of other research medicines in last 1 month.
30. Received or plans to receive an attenuated vaccine within 1 month before or after each study vaccination.
31. Received or plans to receive an inactivated vaccine within 14 days before or after each study vaccination.
32. Current treatment with investigational, authorized, or approved agents for prophylaxis of COVID-19.
33. Have a household contact that has been diagnosed with COVID-19.
34. Current anti-tuberculosis prophylaxis or therapy.
35. Currently receiving treatment for cancer or history of cancer in the last five years (except basal cell carcinoma of the skin and cervical carcinoma in situ).
36. According to the judgement of investigator, various medical, psychological, social or other conditions that could affect the subjects ability to sign informed consent.
37. Assessed by the Investigator to be unable or unwilling to comply with the requirements of the protocol.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2021-02-24 (Actual); Primary Completion 2022-07-11 (Actual); Study Completion 2023-01-09 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Chan Soon - Shiong Institute for Medicine, El Segundo, California
  - Hoag Memorial Hospital Presbyterian, Newport Beach, California

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Cohort 4 - hAd5-S-Fusion+N-ETSD (Suspension for Injection) and hAd5-S-Fusion+N-ETSD (Oral Capsule): For subjects in cohort 4, hAd5-S-Fusion+N-ETSD (Suspension for injection) and hAd5-S-Fusion+N-ETSD (Oral capsule) were administered on day 1 (prime) and hAd5-SFusion+N-ETSD (Oral capsule) were administered on days 15 (boost) and 22 (boost).
  hAd5-S-Fusion+N-ETSD (Suspension for injection): The hAd5-S-Fusion+N-ETSD Vaccine is a human adenovirus serotype 5 (hAd5) vector with E1/E2b/E3 deletions expressing SARS-CoV-2 viral antigen spike fusion protein and nucleocapsid with an enhanced T-cell stimulation domain.
  hAd5-SFusion+ N-ETSD (Oral capsule): The hAd5-S-Fusion+N-ETSD Vaccine is a human adenovirus serotype 5 (hAd5) vector with E1/E2b/E3 deletions expressing SARS-CoV-2 viral antigen spike fusion protein and nucleocapsid with an enhanced T-cell stimulation domain.
Period: Overall Study
Arm/Group | Cohort 1- hAd5-S-Fusion+N-ETSD (Suspension for Injection) and hAd5-SFusion+ N-ETSD (Oral Capsule) | Cohort 2- hAd5-S-Fusion+N-ETSD (Suspension for Injection) and hAd5-SFusion+ N-ETSD (Oral Capsule) | Cohort 3 - hAd5-S-Fusion+N-ETSD (Oral Capsule) | Cohort 4 - hAd5-S-Fusion+N-ETSD (Suspension for Injection) and hAd5-S-Fusion+N-ETSD (Oral Capsule)
Started | 4 | 10 | 10 | 4
Completed | 1 | 10 | 10 | 4
Not Completed | 3 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1- hAd5-S-Fusion+N-ETSD (Suspension for Injection) and hAd5-SFusion+ N-ETSD (Oral Capsule) | Cohort 2- hAd5-S-Fusion+N-ETSD (Suspension for Injection) and hAd5-SFusion+ N-ETSD (Oral Capsule) | Cohort 3 - hAd5-S-Fusion+N-ETSD (Oral Capsule) | Cohort 4 - hAd5-S-Fusion+N-ETSD (Suspension for Injection) and hAd5-S-Fusion+N-ETSD (Oral Capsule) | Total
Number analyzed (Participants) | 4 | 10 | 10 | 4 | 28
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.2 (8.18) | 39.2 (9.67) | 42.2 (10.75) | 44.5 (5.80) | 41.8 (9.24)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 4 | 5 | 2 | 13
  Male | 2 | 6 | 5 | 2 | 15
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 1 | 0 | 3
  Not Hispanic or Latino | 2 | 9 | 9 | 4 | 24
  Unknown or Not Reported | 1 | 0 | 0 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 3 | 1 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 0 | 1 | 0 | 2
  White | 3 | 10 | 5 | 3 | 21
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 1 | 0 | 1
Healthy volunteers with a negative for SARS-CoV-2 test [Count of Participants; unit: Participants] | 4 | 10 | 10 | 4 | 28

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Solicited Local Reactogenicity AEs
Description: Incidence of Solicited Local Treatment-Related Reactogenicity Adverse Events Through 1 Week Post Final Vaccine
Time Frame: 1 week post final vaccine administration
Population: Analysis population is all subjects who received at least one dose of study intervention (safety analysis population)
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1- hAd5-S-Fusion+N-ETSD (Suspension for Injection) and hAd5-SFusion+ N-ETSD (Oral Capsule) | Cohort 2- hAd5-S-Fusion+N-ETSD (Suspension for Injection) and hAd5-SFusion+ N-ETSD (Oral Capsule) | Cohort 3 - hAd5-S-Fusion+N-ETSD (Oral Capsule) | Cohort 4 - hAd5-S-Fusion+N-ETSD (Suspension for Injection) and hAd5-S-Fusion+N-ETSD (Oral Capsule)
Number analyzed (Participants) | 4 | 10 | 10 | 4
Participants | 3 | 8 | 0 | 3

2. Primary Outcome: Incidence of Solicited Systemic Treatment-Related Reactogenicity AEs
Description: Incidence of Solicited Systemic Treatment-Related Reactogenicity Adverse Events Through 1 Week Post Final Vaccine Administration
Time Frame: 1 week post final vaccine administration
Population: Analysis population is all subjects who received at least one dose of study intervention (safety analysis population)
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1- hAd5-S-Fusion+N-ETSD (Suspension for Injection) and hAd5-SFusion+ N-ETSD (Oral Capsule) | Cohort 2- hAd5-S-Fusion+N-ETSD (Suspension for Injection) and hAd5-SFusion+ N-ETSD (Oral Capsule) | Cohort 3 - hAd5-S-Fusion+N-ETSD (Oral Capsule) | Cohort 4 - hAd5-S-Fusion+N-ETSD (Suspension for Injection) and hAd5-S-Fusion+N-ETSD (Oral Capsule)
Number analyzed (Participants) | 4 | 10 | 10 | 4
Participants | 4 | 9 | 7 | 4

3. Primary Outcome: Incidence of Unsolicited AEs
Description: Incidence of Unsolicited AEs Through 1 Week Post Final Vaccine Administration
Time Frame: 1 week post final vaccine administration
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1- hAd5-S-Fusion+N-ETSD (Suspension for Injection) and hAd5-SFusion+ N-ETSD (Oral Capsule) | Cohort 2- hAd5-S-Fusion+N-ETSD (Suspension for Injection) and hAd5-SFusion+ N-ETSD (Oral Capsule) | Cohort 3 - hAd5-S-Fusion+N-ETSD (Oral Capsule) | Cohort 4 - hAd5-S-Fusion+N-ETSD (Suspension for Injection) and hAd5-S-Fusion+N-ETSD (Oral Capsule)
Number analyzed (Participants) | 4 | 10 | 10 | 4
Participants | 2 | 5 | 5 | 3

4. Primary Outcome: Incidence of Unsolicited Treatment-Related AEs
Description: Incidence of Unsolicited Treatment-Related Adverse Events Through 1 Week Post Final Vaccine Administration
Time Frame: 1 week post final vaccine administration
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1- hAd5-S-Fusion+N-ETSD (Suspension for Injection) and hAd5-SFusion+ N-ETSD (Oral Capsule) | Cohort 2- hAd5-S-Fusion+N-ETSD (Suspension for Injection) and hAd5-SFusion+ N-ETSD (Oral Capsule) | Cohort 3 - hAd5-S-Fusion+N-ETSD (Oral Capsule) | Cohort 4 - hAd5-S-Fusion+N-ETSD (Suspension for Injection) and hAd5-S-Fusion+N-ETSD (Oral Capsule)
Number analyzed (Participants) | 4 | 10 | 10 | 4
Participants | 1 | 4 | 4 | 3

5. Primary Outcome: Incidence of Unsolicited AEs
Description: Incidence of Unsolicited Adverse Events Through 30 Days Post Final Vaccine Administration
Time Frame: 30 days post final vaccine
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1- hAd5-S-Fusion+N-ETSD (Suspension for Injection) and hAd5-SFusion+ N-ETSD (Oral Capsule) | Cohort 2- hAd5-S-Fusion+N-ETSD (Suspension for Injection) and hAd5-SFusion+ N-ETSD (Oral Capsule) | Cohort 3 - hAd5-S-Fusion+N-ETSD (Oral Capsule) | Cohort 4 - hAd5-S-Fusion+N-ETSD (Suspension for Injection) and hAd5-S-Fusion+N-ETSD (Oral Capsule)
Number analyzed (Participants) | 4 | 10 | 10 | 4
Participants | 2 | 5 | 5 | 3

6. Primary Outcome: Incidence of Unsolicited Treatment-Related AEs
Description: Incidence of Unsolicited Treatment-Related Adverse Events Through 30 Days Post Final Vaccine Administration
Time Frame: 30 Days Post Final
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1- hAd5-S-Fusion+N-ETSD (Suspension for Injection) and hAd5-SFusion+ N-ETSD (Oral Capsule) | Cohort 2- hAd5-S-Fusion+N-ETSD (Suspension for Injection) and hAd5-SFusion+ N-ETSD (Oral Capsule) | Cohort 3 - hAd5-S-Fusion+N-ETSD (Oral Capsule) | Cohort 4 - hAd5-S-Fusion+N-ETSD (Suspension for Injection) and hAd5-S-Fusion+N-ETSD (Oral Capsule)
Number analyzed (Participants) | 4 | 10 | 10 | 4
Participants | 1 | 4 | 4 | 3

7. Primary Outcome: Incidence of MAAEs
Description: Incidence of Medically Attended Adverse Events Through 6 Months Post Final Vaccine Administration
Time Frame: 6 Months post final vaccine administration
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1- hAd5-S-Fusion+N-ETSD (Suspension for Injection) and hAd5-SFusion+ N-ETSD (Oral Capsule) | Cohort 2- hAd5-S-Fusion+N-ETSD (Suspension for Injection) and hAd5-SFusion+ N-ETSD (Oral Capsule) | Cohort 3 - hAd5-S-Fusion+N-ETSD (Oral Capsule) | Cohort 4 - hAd5-S-Fusion+N-ETSD (Suspension for Injection) and hAd5-S-Fusion+N-ETSD (Oral Capsule)
Number analyzed (Participants) | 4 | 10 | 10 | 4
Participants | 0 | 3 | 4 | 0

8. Primary Outcome: Incidence of Serious AEs
Description: Incidence of Serious Adverse Events Through 6 Months Post- Final Vaccine Administration
Time Frame: 6 Months Post Final Vaccine
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1- hAd5-S-Fusion+N-ETSD (Suspension for Injection) and hAd5-SFusion+ N-ETSD (Oral Capsule) | Cohort 2- hAd5-S-Fusion+N-ETSD (Suspension for Injection) and hAd5-SFusion+ N-ETSD (Oral Capsule) | Cohort 3 - hAd5-S-Fusion+N-ETSD (Oral Capsule) | Cohort 4 - hAd5-S-Fusion+N-ETSD (Suspension for Injection) and hAd5-S-Fusion+N-ETSD (Oral Capsule)
Number analyzed (Participants) | 4 | 10 | 10 | 4
Participants | 0 | 1 | 1 | 0

ADVERSE EVENTS:
Time Frame: Non-serious solicited AEs were to be recorded by the investigator for 7 days after each dose and non-serious unsolicited AEs were to be recorded from the time of first dose of study treatment until 30 days after the last dose of study treatment. All MAAEs, and SAEs were to be recorded by the investigator from the time of first dose of study treatment until 6 months after the last dose of study treatment.
Description: For MAAEs/SAEs that were considered related to study treatment, those events were to be reported at any time regardless of last dose date or end of study visit date.
Groups:
- Group 1:Cohort 1; Group 1: Cohort 2; Group 1:Cohort 3; Group 1:Cohort 4: Solicited Local Reactogenicity Adverse Events Through 1 Week Post Final Vaccine
- Group 2: Cohort 1; Group 2: Cohort 2; Group 2: Cohort 3; Group 2: Cohort 4: Solicited Systemic Reactogenicity Adverse Events Through 1 Week Post Final Vaccine
- Group 3:Cohort 1; Group 3: Cohort 2; Group 3: Cohort 3; Group 3: Cohort 4: Unsolicited Adverse Events Through 1 Week Post Final Vaccine Administration
- Group 4: Cohort 1; Group 4: Cohort 2; Group 4: Cohort 3; Group 4: Cohort 4: Unsolicited Treatment-Related Adverse Events Through 1 Week Post Final Vaccine Administration
- Group 5: Cohort 1; Group 5:Cohort 2; Group 5: Cohort 3; Group 5: Cohort 4: Unsolicited Adverse Events Through 30 Days Post Final Vaccine Administration
- Group 6: Cohort 1; Group 6: Cohort 2; Group 6: Cohort 3; Group 6: Cohort 4: Unsolicited Treatment-Related Adverse Events Through 30 Days Post Final Vaccine Administration
- Group 7: Cohort 1; Group 7: Cohort 2; Group 7:Cohort 3; Group 7: Cohort 4: Incidence of Medically Attended Adverse Events Through 6 Months Post Final Vaccine Administration
Arm/Group | Group 1:Cohort 1 | Group 1: Cohort 2 | Group 1:Cohort 3 | Group 1:Cohort 4 | Group 2: Cohort 1 | Group 2: Cohort 2 | Group 2: Cohort 3 | Group 2: Cohort 4 | Group 3:Cohort 1 | Group 3: Cohort 2 | Group 3: Cohort 3 | Group 3: Cohort 4 | Group 4: Cohort 1 | Group 4: Cohort 2 | Group 4: Cohort 3 | Group 4: Cohort 4 | Group 5: Cohort 1 | Group 5:Cohort 2 | Group 5: Cohort 3 | Group 5: Cohort 4 | Group 6: Cohort 1 | Group 6: Cohort 2 | Group 6: Cohort 3 | Group 6: Cohort 4 | Group 7: Cohort 1 | Group 7: Cohort 2 | Group 7:Cohort 3 | Group 7: Cohort 4
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/10 | 0/10 | 0/4 | 0/4 | 0/10 | 0/10 | 0/4 | 0/4 | 0/10 | 0/10 | 0/4 | 0/4 | 0/10 | 0/10 | 0/4 | 0/4 | 0/10 | 0/10 | 0/4 | 0/4 | 0/10 | 0/10 | 0/4 | 0/4 | 0/10 | 0/10 | 0/4
Serious Adverse Events (participants affected / at risk) | 0/4 | 1/10 | 1/10 | 0/4 | 0/4 | 0/10 | 0/10 | 0/4 | 0/4 | 0/10 | 0/10 | 0/4 | 0/4 | 0/10 | 0/10 | 0/4 | 0/4 | 0/10 | 0/10 | 0/4 | 0/4 | 0/10 | 0/10 | 0/4 | 0/4 | 0/10 | 0/10 | 0/4
Other Adverse Events (participants affected / at risk) | 3/4 | 8/10 | 0/10 | 3/4 | 4/4 | 9/10 | 7/10 | 4/4 | 2/4 | 5/10 | 5/10 | 3/4 | 1/4 | 4/10 | 4/10 | 3/4 | 2/4 | 5/10 | 5/10 | 3/4 | 1/4 | 4/10 | 4/10 | 3/4 | 0/4 | 3/10 | 4/10 | 0/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Group 1:Cohort 1 (N=4) | Group 1: Cohort 2 (N=10) | Group 1:Cohort 3 (N=10) | Group 1:Cohort 4 (N=4) | Group 2: Cohort 1 (N=4) | Group 2: Cohort 2 (N=10) | Group 2: Cohort 3 (N=10) | Group 2: Cohort 4 (N=4) | Group 3:Cohort 1 (N=4) | Group 3: Cohort 2 (N=10) | Group 3: Cohort 3 (N=10) | Group 3: Cohort 4 (N=4) | Group 4: Cohort 1 (N=4) | Group 4: Cohort 2 (N=10) | Group 4: Cohort 3 (N=10) | Group 4: Cohort 4 (N=4) | Group 5: Cohort 1 (N=4) | Group 5:Cohort 2 (N=10) | Group 5: Cohort 3 (N=10) | Group 5: Cohort 4 (N=4) | Group 6: Cohort 1 (N=4) | Group 6: Cohort 2 (N=10) | Group 6: Cohort 3 (N=10) | Group 6: Cohort 4 (N=4) | Group 7: Cohort 1 (N=4) | Group 7: Cohort 2 (N=10) | Group 7:Cohort 3 (N=10) | Group 7: Cohort 4 (N=4)
Diverticulitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA
Radius fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Group 1:Cohort 1 (N=4) | Group 1: Cohort 2 (N=10) | Group 1:Cohort 3 (N=10) | Group 1:Cohort 4 (N=4) | Group 2: Cohort 1 (N=4) | Group 2: Cohort 2 (N=10) | Group 2: Cohort 3 (N=10) | Group 2: Cohort 4 (N=4) | Group 3:Cohort 1 (N=4) | Group 3: Cohort 2 (N=10) | Group 3: Cohort 3 (N=10) | Group 3: Cohort 4 (N=4) | Group 4: Cohort 1 (N=4) | Group 4: Cohort 2 (N=10) | Group 4: Cohort 3 (N=10) | Group 4: Cohort 4 (N=4) | Group 5: Cohort 1 (N=4) | Group 5:Cohort 2 (N=10) | Group 5: Cohort 3 (N=10) | Group 5: Cohort 4 (N=4) | Group 6: Cohort 1 (N=4) | Group 6: Cohort 2 (N=10) | Group 6: Cohort 3 (N=10) | Group 6: Cohort 4 (N=4) | Group 7: Cohort 1 (N=4) | Group 7: Cohort 2 (N=10) | Group 7:Cohort 3 (N=10) | Group 7: Cohort 4 (N=4)
Injection site pain (General disorders) | 3 | 6 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | 0 | 0 | 0
Injection site erythema (General disorders) | 3 | 3 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | NA | 0 | 0 | 0
Injection site pruritus (General disorders) | 2 | 3 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | NA | 0 | 0 | 0
Injection site reaction (General disorders) | 1 | 4 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | 0 | 0 | 0
Injection site swelling (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | 0 | 0 | 0
Fatigue (General disorders) | 0 | 0 | 0 | 0 | 4 | 8 | 6 | 4 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Chills (General disorders) | 0 | 0 | 0 | 0 | 2 | 4 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nausea (General disorders) | 0 | 0 | 0 | 0 | 2 | 7 | 4 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 4 | 6 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 3 | 2 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal discomfort (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 0 | 0 | 0 | 0 | 2 | 8 | 5 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 5 | 4 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Feeling abnormal (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 1 | 0 | 2 | 1 | 1 | 0 | 2 | 1 | 1 | 0 | 2 | 1 | 1 | 0 | 0 | 0 | 0
Feeling hot (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Injection site induration (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Non-cardiac chest pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pyrexia (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Swelling Face (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Vessel puncture site pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dysgeusia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hypoaesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Migraine (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Paraesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Flatulence (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 2 | 1 | 0 | 0 | 0 | NA
Hyperaesthesia teeth (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Paraesthesia oral (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 1 | 1 | 0 | 0 | 2 | 1 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 1 | 1 | 0 | 1 | 1 | 1 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Ear discomfort (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ear pain (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Tinnitus (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Back Pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Palpitations (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Eye discharge (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ocular discomfort (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Dysuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hot flush (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Throat tightness (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Forearm Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Radius Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Ehlers-Danlos syndrome (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Gastric polyps (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Gastritis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Diverticulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Anxiety (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Acne (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0

LIMITATIONS AND CAVEATS:
The study was terminated early due to low enrollment.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-03-31): https://cdn.clinicaltrials.gov/large-docs/68/NCT04732468/Prot_SAP_000.pdf